CLINICAL TRIAL: NCT07254364
Title: Advancing Precision Nutrition: Wearable Technology for Noninvasive Insulin Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 105-Sweat
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Insulin Response

STUDY DESIGN:
Intervention Model Description: Individual response to a standardized liquid nutrition meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized liquid meal drink (Experimental): We will provide a standardized drink consisting of whey, maltodextrin and sunflower oil, flavored using vanilla sugar-free instant pudding.
  Interventions: Other: Standardized meal

INTERVENTIONS:
Other: Standardized meal — We will use Whey powder (60g) as protein, Maltodextrin (Polycose; 170g) as carbohydrate, and Sunflower Oil (48g) as the fat source. The meal is mixed and flavored using vanilla sugar-free instant pudding.

SUMMARY:
Noninvasively monitoring insulin is crucial for advancing precision nutrition and promoting healthy living by enabling a deeper understanding of individual metabolic responses to dietary intake. Insulin is a key regulator of blood sugar and energy metabolism, and its dysregulation is linked to conditions such as diabetes, obesity, and metabolic syndrome. By noninvasively tracking insulin levels, individuals can gain real-time insights into how their body processes different foods, allowing for the personalization of diets to optimize metabolic health, manage weight, and reduce disease risk. This approach also empowers proactive lifestyle adjustments to maintain insulin sensitivity, improve glycemic control, and enhance overall well-being. Decentralized insulin quantification in biofluids, including saliva and serum, based on lateral flow assay or electrochemical sensor has been reported. However, these approaches have poor sensitivity and fail to quantify insulin with a high temporal resolution.

DETAILED DESCRIPTION:
The goal of the proposed research is to develop a wearable device that can directly stimulate sweat secretion and rapidly quantify the concentration of insulin in sweat. In stark contrast to a blood draw and subsequent insulin quantification in a clinical lab, the envisioned wearable sweat sensor can noninvasively and rapidly quantify insulin at any desired time at home. This study will validate the performance of the wearable devices for in situ quantification of insulin in sweat and determine the concentration correlation between sweat, dermal interstitial fluid, and blood.

The study will take place at the research facility of the Center for Translational Research on Aging and Longevity (CTRAL), Texas A&M University located in the Human Clinical Research Building) affiliated with Texas A&M University. Some study procedures (e.g., body composition) may be skipped if completed within the past 3 months at CTRAL. All data will be recorded in Case Report Form and stored in the Research Electronic Data Capturing (REDCap) System.

Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight, height, and body composition by Dualenergy X-ray absorptiometry (DXA) will be measured. In addition, The SixMinute Walk Test (6MWT) and skeletal muscle function tests will be assessed at the end of each screening visit. Questionnaires about your overall health and well-being will also be completed. The study visit will begin with vital signs. Before administration of the feeding or the tracer solution, baseline blood will be collected for measurement of the natural enrichment of metabolites. The research nurse will place a catheter (small, flexible, plastic tube) in a vein of the arm or hand. The hand will be placed in a warmed box to increase blood flow. There will be a device with electrodes used to generate and collect sweat on your forearm. Once sweat collection is started, we will also apply a microneedle patch to the forearm of the subject for 5-30 minutes duration. Microneedle patches (sensors) are small flexible sticker-like devices. They will be applied to the skin using a small spring loaded applicator to measure the chemical analytes in the dermal interstitial fluids. After 2 hours of baseline biological samples of sweat, dermal interstitial fluid, and blood have been collected, we will provide a standardized meal as a liquid drink consisting of whey, maltodextrin and sunflower oil, flavored using vanilla sugar-free instant pudding. Biological sampling will continue to occur for the following 5 hours.

ELIGIBILITY:
Inclusion criteria:

* Age

  * 18-30 years old
  * 50-90 years old
* BMI between 22 and 35 kg/m2
* Ability to walk, sit down, and stand up (independently or with a walking assistance device)
* Willingness to lay supine in bed for up to 9 hours
* Willingness and ability to comply with the protocol

Exclusion criteria

* Known allergy to any of the components of the meal or agents used for the application of the devices

  * Sunflower oil
  * Maltodextrin
  * Whey protein
  * Pilocarpine solutions
* Established diagnosis and active treatment of chronic disease: insulin-dependent diabetes, active malignancy, heart failure, kidney disease, liver disease, HIV/AIDS, asthma (moderate to severe), Hep (A, B, or C)
* History of untreated metabolic disease including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Active dependence on alcohol or drugs
* Use of a short course of oral corticosteroids within 4 weeks preceding study day
* Current use of long-term oral corticosteroids
* Presence of fever within the last 3 days
* Planned elective surgery requiring 2 or more days of hospitalization during the entire study
* (Possible) pregnancy (confirmed via urine pregnancy test for females 18-30 years)
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject
* Any condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of protein biomarkers | up to 9 hours, 1 day
  Time-varying plasma insulin concentrations and correlation between sweat and dermal interstitial fluid.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT07254364/ICF_000.pdf